CLINICAL TRIAL: NCT02567019
Title: Immunoregulation of Periodontal Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-A00882-47
Record Dates: First submitted 2015-08-31; First posted 2015-10-02 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Parodontosis
MeSH Terms: conditions — Periodontal Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- periodontal diseases (Experimental): blood samples will be done for patients suffering of periodontal diseases
  Interventions: Other: blood samples
- healthy volunteers (Active Comparator): blood samples will be done for healthy volunteers
  Interventions: Other: blood samples

INTERVENTIONS:
Other: blood samples — blood samples will be done for patients patients suffering of periodontal diseases and healthy volunteers

SUMMARY:
Periodontal diseases are a group of diseases that affect 15% of the population and in the absence of treatment causes tooth loss. Periodontal lesions are characterized mainly by strong inflammation and hyper-vascularization. Search in blood cells and inflammatory markers attempts to explain the etiological-pathogenetic mechanisms. Innate immunity can be assessed by qualitative and quantitative analysis of blood phagocytes, natural killer cells, complement, proteins of inflammation and cytokines. Current data from the literature on this subject give contradictory results and the comparison of studies are difficult because the diversity of the populations studied, evaluated cells and the methods used. The aim of the study was to evaluate the innate immunity of patients with periodontal disease and compare it with a group of patients without periodontal disease.

DETAILED DESCRIPTION:
Periodontal diseases are a group of diseases that affect 15% of the population and in the absence of treatment causes tooth loss. Periodontal lesions are characterized mainly by strong inflammation and hyper-vascularization. Search in blood cells and inflammatory markers attempts to explain the etiological-pathogenetic mechanisms. Innate immunity can be assessed by qualitative and quantitative analysis of blood phagocytes, natural killer cells, complement, proteins of inflammation and cytokines. Current data from the literature on this subject give contradictory results and the comparison of studies are difficult because the diversity of the populations studied, evaluated cells and the methods used. The aim of the study was to evaluate the innate immunity of patients with periodontal disease and compare it with a group of patients without periodontal disease. The previous conclusions of study focused on the difference in the general immunological parameters in healthy patients and patients suffering from periodontal disease, current advances in immunology have helped to develop new markers on functional status of blood phagocytes all through their anti-microbial action. The adhesion, migration, phagocytosis and bactericidal capacity are assessed and quantified using recognized tests and practiced regularly in analytical laboratory. The identification of altered immunological parameters in patients with periodontal disease would better understand the natural history of these diseases and may lead to new diagnostic criteria, prognostic and therapeutic.

In practice, the project brings together immunological skills (functional analysis of cells and membrane markers) and dental (patient selection and diagnosis of periodontal disease) for further testing applicable to many patients likely to develop periodontal disease.

ELIGIBILITY:
Inclusion Criteria:

For periodontal subjects

* At least present 20 teeth on the dental arches
* Presence of periodontal deep pockets = 4 mm measured by means of a periodontal probe increased in millimeters and raised on at least 30 % of the dental surfaces (proximal, vestibular and Palatine or lingual) present teeth on the dental arches.

For healthy volunteers : absence of periodontal deep pockets

Exclusion Criteria:

* pathologies or treatments whom could affect the immunological parameters for the both arms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
% phagocytes cells of blood | 1 year
  Identification of altered immunological parameters in patients with periodontal disease

CONTACTS AND LOCATIONS:
Overall Officials: Virgine MONNET CORTI, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France